CLINICAL TRIAL: NCT03421080
Title: Does Providing a Brief Internet Intervention for Hazardous Alcohol Use to People Seeking Online Help for Depression Reduce Both Alcohol Use and Depression Symptoms Among Participants With These Co-occurring Disorders? Randomized Controlled Trial
Brief Title: Brief Internet Intervention for Hazardous Alcohol Use to People Seeking Online Help for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, John Cunningham, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 064/2017
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Depression; Problem Drinking
MeSH Terms: conditions — Depression; Alcoholism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MoodGYM Only (Active Comparator): The MoodGYM only Internet intervention will consist of a popular, automated, self-help cognitive behavioral therapy program for depression comprising five modules to be completed over five weeks and an online workbook incorporating 29 exercises. A series of published research trials has shown MoodGYM to be effective in reducing depressive symptoms in users in a range of settings (e.g., schools, universities, Lifeline suicide prevention, U.K. NHS Choices online), for different aspects of the mental health service spectrum (e.g., prevention vs treatment), and different age groups (adults, adolescents).
  Interventions: Behavioral: MoodGYM
- MoodGYM + CYD (Experimental): The MoodGYM + CYD intervention condition will consist of the MoodGYM only intervention and an online intervention providing feedback on quantity and frequency of drinking, severity of hazardous drinking, and provides recommendations for safe levels of alcohol consumption (Check Your Drinking - CYD). The CYD Final Report will be provided as part of the participant's MoodDYM dashboard.
  Interventions: Behavioral: MoodGYM; Behavioral: Check Your Drinking

INTERVENTIONS:
Behavioral: MoodGYM — The MoodGYM Internet intervention will employ the latest version of MoodGYM (Mark 4) which has been updated to support mobile devices. The core design and function of the program has not been altered. A major focus of this intervention is to provide individuals with behavioral and cognitive strategies to improve depression symptoms.
Behavioral: Check Your Drinking — Internet intervention designed to assess and provide feedback on hazardous alcohol use. The CYD has been subjected to seven randomized trials from two independent research groups, all of which displayed a significant impact of the CYD to reduce hazardous alcohol consumption compared to controls.
  Arms: MoodGYM + CYD

SUMMARY:
Hazardous alcohol consumption is common among people suffering from depression. There are effective Internet interventions that target hazardous alcohol consumption or depression separately but none that combine these online interventions without the involvement of a therapist. This study aims to evaluate the effects of combining an Internet intervention targeting hazardous alcohol consumption with one for depression on drinking and depressive symptoms.

DETAILED DESCRIPTION:
A double-blinded, parallel group randomized controlled trial will be used. Participants with current depression who also drink in a hazardous fashion (N=986) will be recruited for a study to 'help improve an online intervention for depression.' Participants will be assigned, by chance, to receive MoodGYM or to receive MoodGYM plus a brief Internet intervention for hazardous alcohol consumption - Check Your Drinking (CYD). Participants will be contacted 3- and 6-months after receiving the interventions to assess changes in drinking and depression status. It is predicted that participants receiving the CYD intervention in addition to MoodGYM will reduce their alcohol consumption to a greater extent than those who just received MoodGYM. Further predictions include the impact of receiving Check Your Drinking on improvements in depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or over
* score 10 or more on the Patient Health Questionnaire (PHQ-9)
* score 8 or more on the Alcohol Use Disorder Identification Test (AUDIT)

Exclusion Criteria:

* current suicidal ideation on the PHQ-9

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 988 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
Number of drinks in a typical week | 3 and 6 months
  Change in number of drinks in a typical week from baseline

SECONDARY OUTCOMES:
CES-D | 3 and 6 months
  Change in depressive symptoms using the Centre for Epidemiological Studies Depression scale (CES-D) from baseline. Total score range from zero to 60 with higher scores indicating more symptomatology.
AUDIT-C | 3 and 6 months
  Change in AUDIT-C score (consumption subscale from the AUDIT) from baseline
Alcohol consequences | 3 and 6 months
  Change in number of alcohol consequences from baseline

OTHER OUTCOMES:
Health related quality of life | 3 and 6 months
  Measure changes in health related quality of life from baseline (EUROHIS-QoL8)

CONTACTS AND LOCATIONS:
Overall Officials: John A Cunningham, Ph.D., Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cunningham JA, Godinho A, Hendershot CS, Kay-Lambkin F, Neighbors C, Griffiths KM, Schell C. Randomized controlled trial of online interventions for co-occurring depression and hazardous alcohol consumption: Primary outcome results. Internet Interv. 2021 Nov 2;26:100477. doi: 10.1016/j.invent.2021.100477. eCollection 2021 Dec. PMID 34786350
- [Derived] Godinho A, Schell C, Cunningham JA. Falling between the cracks: The effect of using different levels of suicide risk exclusion criteria on sample characteristics when recruiting for an online intervention for depression. Suicide Life Threat Behav. 2021 Aug;51(4):736-740. doi: 10.1111/sltb.12761. Epub 2021 May 7. PMID 33961291
- [Derived] Cunningham JA, Hendershot CS, Kay-Lambkin F, Neighbors C, Griffiths KM, Bennett K, Bennett A, Godinho A, Schell C. Does providing a brief internet intervention for hazardous alcohol use to people seeking online help for depression reduce both alcohol use and depression symptoms among participants with these co-occurring disorders? Study protocol for a randomised controlled trial. BMJ Open. 2018 Jul 19;8(7):e022412. doi: 10.1136/bmjopen-2018-022412. PMID 30030322
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre — http://www.camh.ca/en/research